CLINICAL TRIAL: NCT00380250
Title: Phase 3, 12-Week, Multicenter, Double-Blind, Randomized, Efficacy and Safety Study of Lubiprostone for the Treatment of Irritable Bowel Syndrome With Constipation
Brief Title: Efficacy and Safety of Lubiprostone in Patients With Irritable Bowel Syndrome With Constipation
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sucampo Pharma Americas, LLC (Industry)
Collaborators: Takeda (Industry)
Responsible Party: Sponsor
Organization: Mallinckrodt (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0211SIB-0431
Record Dates: First submitted 2006-09-21; First posted 2006-09-25 (Estimated); Results first posted 2014-02-11 (Estimated); Last update posted 2019-11-15 (Actual); Status verified 2014-01

CONDITIONS: Irritable Bowel Syndrome With Constipation
MeSH Terms: interventions — Lubiprostone

ARMS (2):
- Lubiprostone (Experimental): 8 mcg capsule twice daily (BID)
  Interventions: Drug: Lubiprostone
- Placebo (Placebo Comparator): Matching placebo capsule twice daily (BID)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Lubiprostone
  Arms: Lubiprostone
Drug: Placebo
  Arms: Placebo

SUMMARY:
The primary purpose of this study is to evaluate the efficacy and safety of administration of lubiprostone in patients with irritable bowel syndrome with constipation.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age and older
* Stable fiber therapy
* Normal colonoscopy/sigmoidoscopy
* Able to refrain from use of medications known to treat or associated with constipation symptoms
* Experiences abdominal discomfort/pain associated with bowel movements
* Reports decreased bowel movement frequency and/or other symptoms associated with constipation

Exclusion Criteria:

* Diarrhea-predominant or alternating (diarrhea and constipation cycling) irritable bowel syndrome (IBS), or constipation other than that associated with IBS
* Open gastrointestinal or abdominal surgery prior to IBS onset
* Organic bowel disorder, mechanical bowel obstruction, pseudo-obstruction, unexplained weight loss or rectal bleeding
* Uncontrolled cardiovascular, liver or lung disease, neurologic or psychiatric disorder, other systemic disease, or abnormal laboratory tests per investigator discretion
* If female, is currently pregnant or nursing, or plans to become pregnant or nurse during the clinical study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 590 (Actual)
Dates: Start 2005-05; Study Completion 2006-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, MD, Study Director — Sucampo Pharmaceuticals, Inc.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Drossman DA, Chey WD, Johanson JF, Fass R, Scott C, Panas R, Ueno R. Clinical trial: lubiprostone in patients with constipation-associated irritable bowel syndrome--results of two randomized, placebo-controlled studies. Aliment Pharmacol Ther. 2009 Feb 1;29(3):329-41. doi: 10.1111/j.1365-2036.2008.03881.x. Epub 2008 Nov 4. PMID 19006537

RESULTS

PARTICIPANT FLOW:
Recruitment Details: First subject entered 5/12/05; Last subject observation 7/18/08; Multicenter study performed at 65 study sites/centers across the US
Pre-assignment Details: Subjects were enrolled after an up to 4 week screening period to meet inclusion/exclusion criteria and randomized on Day 0
Groups:
- Lubiprostone Study Period I: Subjects who received active drug
- Placebo Study Period I: Subjects who received placebo
Period: Overall Study
Arm/Group | Lubiprostone Study Period I | Placebo Study Period I
Started | 396 | 194
Completed | 297 | 139
Not Completed | 99 | 55
Not completed — Withdrawal by Subject | 39 | 28
Not completed — Adverse Event | 20 | 9
Not completed — Lack of Efficacy | 10 | 8
Not completed — Protocol Violation | 15 | 5
Not completed — Lost to Follow-up | 14 | 5
Not completed — Physician Decision | 1 | 0

BASELINE CHARACTERISTICS:
Population: The Baseline participants data is taken from the intent to treat(ITT) population Whereas the Participant flow data is for all randomized subjects.
Groups:
- Total: Total of all reporting groups
Arm/Group | Lubiprostone Study Period I | Placebo Study Period I | Total
Number analyzed (Participants) | 390 | 193 | 583
Age, Continuous [Mean (Full Range); unit: years] | 46.7 [19 to 83] | 48.1 [20 to 85] | 47.2 [19 to 85]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 355 | 180 | 535
  Male | 35 | 13 | 48
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 53 | 29 | 82
  White | 336 | 160 | 496
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 3 | 3
Height [Mean (Standard Deviation); unit: Inches] | 64.9 (2.9) | 64.8 (3.09) | 64.9 (2.96)

OUTCOME MEASURES:

1. Secondary Outcome: Month 1 Spontaneous Bowel Movement (SBM) Frequency Rates Change From Baseline
Description: SBMs are any bowel movement not associated with rescue medication use.
Time Frame: Change from baseline for month 1
Population: ITT with LOCF
Measure: Mean (Standard Deviation); unit: SBM/week
Arm/Group | Lubiprostone Study Period I | Placebo Study Period I
Number analyzed (Participants) | 390 | 193
SBM/week | 1.54 (2.462) | 1.21 (2.286)
Statistical Analysis 1: Comparison: Lubiprostone Study Period I vs Placebo Study Period I; Test type: Superiority or Other; p = 0.117, van Elteren nonparametric test; Adjusted for center

2. Secondary Outcome: Month 1 Stool Consistency Change From Baseline
Description: 0 = Very loose (watery), 1 = Loose, 2 = Normal, 3 = Hard, 4 = Very hard (little balls)
Time Frame: Change from baseline for month 1
Population: ITT with LOCF
Measure: Mean (Standard Deviation); unit: Scale score
Arm/Group | Lubiprostone Study Period I | Placebo Study Period I
Number analyzed (Participants) | 390 | 193
Scale score | -0.51 (0.690) | -0.33 (0.626)
Statistical Analysis 1: Comparison: Lubiprostone Study Period I vs Placebo Study Period I; Test type: Superiority or Other; p = 0.006, van Elteren nonparametric test; Adjusted for center

3. Secondary Outcome: Month 1 Bowel Straining Change From Baseline
Description: 0 = Absent,1 = Mild, 2 = Moderate, 3 = Severe, and 4 = Very Severe
Time Frame: Change from baseline for month 1
Population: ITT with LOCF
Measure: Mean (Standard Deviation); unit: Scale score
Arm/Group | Lubiprostone Study Period I | Placebo Study Period I
Number analyzed (Participants) | 390 | 193
Scale score | -0.53 (0.739) | -0.36 (0.694)
Statistical Analysis 1: Comparison: Lubiprostone Study Period I vs Placebo Study Period I; Test type: Superiority or Other; p = 0.050, van Elteren nonparametric test; Adjusted for center

4. Secondary Outcome: Month 1 Constipation Severity Change From Baseline
Description: 0 = Absent, 1 = Mild, 2 = Moderate, 3 = Severe, and 4 = Very Severe
Time Frame: Change from baseline at 28 days
Population: ITT with LOCF
Measure: Mean (Standard Deviation); unit: Scale score
Arm/Group | Lubiprostone Study Period I | Placebo Study Period I
Number analyzed (Participants) | 390 | 193
Scale score | -0.41 (0.602) | -0.29 (0.568)
Statistical Analysis 1: Comparison: Lubiprostone Study Period I vs Placebo Study Period I; Test type: Superiority or Other; p = 0.159, van Elteren nonparametric test; Adjusted for center

5. Secondary Outcome: Month 1 Symptom Relief
Description: Significantly worse = -3; Moderately worse = -2; A little bit worse = -1; Unchanged = 0; A little bit relieved=1; Moderately relieved=2; Significantly relieved = 3
Time Frame: Change from baseline for month 1
Population: ITT with LOCF
Measure: Mean (Standard Deviation); unit: Scale score
Arm/Group | Lubiprostone Study Period I | Placebo Study Period I
Number analyzed (Participants) | 390 | 193
Scale score | 0.66 (1.212) | 0.57 (1.088)
Statistical Analysis 1: Comparison: Lubiprostone Study Period I vs Placebo Study Period I; Test type: Superiority or Other; p = 0.378, Cochran-Mantel-Haenszel; Stratified by pooled center

6. Secondary Outcome: Quality of Life Change From Baseline
Description: Irritable Bowel Syndrome Quality of Life (IBS-QOL) questionnaire included 34 questions with 5 possible responses yielding the following sub-categories: dysphoria, interference with activity, body image, health worry, food avoidance, social reaction, sexual, and relationship Results range from 34 (low) to 100 (high); meaningful clinical improvement=14 point increase
Time Frame: Change from baseline at 12 weeks
Population: ITT without LOCF
Measure: Mean (Standard Deviation); unit: Scale score
Arm/Group | Lubiprostone Study Period I | Placebo Study Period I
Number analyzed (Participants) | 390 | 193
Scale score | 16.7 (17.36) | 16.8 (19.72)
Statistical Analysis 1: Comparison: Lubiprostone Study Period I vs Placebo Study Period I; Test type: Superiority or Other; p = 0.588, ANCOVA; Adjusted for clinical site

7. Primary Outcome: Overall Responder Rate
Description: Monthly responder: >=Moderately relieved symptoms 4 weeks/month or Significantly relieved >= 2 weeks/month IF:
  Rescue med use did not increase during the month; AND did not discontinue during the month for lack of efficacy; AND no Moderately worse or Significantly worse response in month.
  Overall responder: responder for at least 2/3 months
Time Frame: 12 weeks
Population: Intent-to-treat (ITT) without Last Observation Carried Forward (LOCF)
Measure: Number; unit: percentage of participants
Arm/Group | Lubiprostone Study Period I | Placebo Study Period I
Number analyzed (Participants) | 390 | 193
percentage of participants | 13.8 | 7.8
Statistical Analysis 1: Comparison: Lubiprostone Study Period I vs Placebo Study Period I; 90% statistical power to detect 70.6% improvement in response with lubiprostone; Test type: Superiority or Other; p = 0.029, Cochran-Mantel-Haenszel — No adjustment; Stratified by pooled center, used to test the null hypothesis of equal rates between the 2 groups vs. the alternate hypothesis of non-equality

8. Secondary Outcome: Month 2 Responder Rate
Description: Monthly responder: >=Moderately relieved symptoms 4 weeks/month or Significantly relieved >= 2 weeks/month IF:
  Rescue med use did not increase during the month; AND did not discontinue during the month for lack of efficacy; AND no Moderately worse or Significantly worse response in month.
Time Frame: month 2 (28 days)
Population: ITT without LOCF
Measure: Number; unit: percent of participants
Arm/Group | Lubiprostone Study Period I | Placebo Study Period I
Number analyzed (Participants) | 390 | 193
percent of participants | 15.9 | 9.3
Statistical Analysis 1: Comparison: Lubiprostone Study Period I vs Placebo Study Period I; Test type: Superiority or Other; p = 0.028, Cochran-Mantel-Haenszel — Sequential closed testing procedures were employed; [statistical method as in outcome 7, analysis 1]

9. Secondary Outcome: Month 3 Responder Rate
Description: Symptoms >= Moderately relieved for 4 weeks/month or Significantly relieved for >=2 weeks/month AND:
  1. Rescue medication use does not increase during the month as compared to baseline;
  2. No discontinuation during the month due to lack of efficacy;AND
  3. No ratings during the month of Moderately worse or Significantly worse.
Time Frame: month 3 (28 days)
Population: ITT without LOCF
Measure: Number; unit: percent of participants
Arm/Group | Lubiprostone Study Period I | Placebo Study Period I
Number analyzed (Participants) | 390 | 193
percent of participants | 15.9 | 10.4
Statistical Analysis 1: Comparison: Lubiprostone Study Period I vs Placebo Study Period I; Test type: Superiority or Other; p = 0.069, Cochran-Mantel-Haenszel — Sequential closed testing procedures were employed; [statistical method as in outcome 7, analysis 1]

10. Secondary Outcome: Month 1 Responder Rate
Description: as for outcome 9
Time Frame: month 1 (28 days)
Population: ITT without LOCF
Measure: Number; unit: percent of participants
Arm/Group | Lubiprostone Study Period I | Placebo Study Period I
Number analyzed (Participants) | 390 | 193
percent of participants | 10.0 | 6.2
Statistical Analysis 1: Comparison: Lubiprostone Study Period I vs Placebo Study Period I; Test type: Superiority or Other; p = 0.098, Cochran-Mantel-Haenszel — Sequential closed testing procedures were employed; [statistical method as in outcome 7, analysis 1]

11. Secondary Outcome: Month 2 Abdominal Bloating Change From Baseline
Description: 0 = Absent, 1 = Mild, 2 = Moderate, 3 = Severe, and 4 = Very Severe
Time Frame: Change from baseline for month 2
Population: ITT with LOCF
Measure: Mean (Standard Deviation); unit: Scale score
Arm/Group | Lubiprostone Study Period I | Placebo Study Period I
Number analyzed (Participants) | 390 | 193
Scale score | -0.42 (0.693) | -0.35 (0.621)
Statistical Analysis 1: Comparison: Lubiprostone Study Period I vs Placebo Study Period I; Test type: Superiority or Other; p = 0.286, van Elteren nonparametric test; Adjusted for center

12. Secondary Outcome: Month 3 Abdominal Bloating Change From Baseline
Description: 0 = Absent, 1 = Mild, 2 = Moderate, 3 = Severe, and 4 = Very Severe
Time Frame: Change from baseline for month 3
Population: ITT with LOCF
Measure: Mean (Standard Deviation); unit: Scale score
Arm/Group | Lubiprostone Study Period I | Placebo Study Period I
Number analyzed (Participants) | 390 | 193
Scale score | -0.43 (0.734) | -0.37 (0.693)
Statistical Analysis 1: Comparison: Lubiprostone Study Period I vs Placebo Study Period I; Test type: Superiority or Other; p = 0.337, van Elteren nonparametric test; Adjusted for center

13. Secondary Outcome: Month 2 Spontaneous Bowel Movement Frequency Rates Change From Baseline
Description: Any bowel movement not associated with rescue medication use
Time Frame: Change from baseline for month 2
Population: ITT with LOCF
Measure: Mean (Standard Deviation); unit: SBM/week
Arm/Group | Lubiprostone Study Period I | Placebo Study Period I
Number analyzed (Participants) | 390 | 193
SBM/week | 1.59 (2.795) | 1.41 (2.587)
Statistical Analysis 1: Comparison: Lubiprostone Study Period I vs Placebo Study Period I; Test type: Superiority or Other; p = 0.334, van Elteren nonparametric test; Adjusted for center

14. Secondary Outcome: Month 3 Spontaneous Bowel Movement Frequency Rates Change From Baseline
Description: Any bowel movement not associated with rescue medication use
Time Frame: Change from baseline for month 3
Population: ITT with LOCF
Measure: Mean (Standard Deviation); unit: SBM/week
Arm/Group | Lubiprostone Study Period I | Placebo Study Period I
Number analyzed (Participants) | 390 | 193
SBM/week | 1.51 (2.990) | 1.39 (2.851)
Statistical Analysis 1: Comparison: Lubiprostone Study Period I vs Placebo Study Period I; Test type: Superiority or Other; p = 0.242, van Elteren nonparametric test; Adjusted for center

15. Secondary Outcome: Month 2 Stool Consistency Change From Baseline
Description: 0 = Very loose (watery), 1 = Loose, 2 = Normal, 3 = Hard, 4 = Very hard (little balls)
Time Frame: Change from baseline for month 2
Population: ITT with LOCF
Measure: Mean (Standard Deviation); unit: Scale score
Arm/Group | Lubiprostone Study Period I | Placebo Study Period I
Number analyzed (Participants) | 390 | 193
Scale score | -0.53 (0.756) | -0.38 (0.658)
Statistical Analysis 1: Comparison: Lubiprostone Study Period I vs Placebo Study Period I; Test type: Superiority or Other; p = 0.030, van Elteren nonparametric test; Adjusted for center

16. Secondary Outcome: Month 3 Stool Consistency Change From Baseline
Description: 0 = Very loose (watery), 1 = Loose, 2 = Normal, 3 = Hard, 4 = Very hard (little balls)
Time Frame: Change from baseline for month 3
Population: ITT with LOCF
Measure: Mean (Standard Deviation); unit: Scale score
Arm/Group | Lubiprostone Study Period I | Placebo Study Period I
Number analyzed (Participants) | 390 | 193
Scale score | -0.52 (0.725) | -0.41 (0.696)
Statistical Analysis 1: Comparison: Lubiprostone Study Period I vs Placebo Study Period I; Test type: Superiority or Other; p = 0.130, van Elteren nonparametric test; Adjusted for center

17. Secondary Outcome: Month 2 Bowel Straining Change From Baseline
Description: 0 = Absent,1 = Mild, 2 = Moderate, 3 = Severe, and 4 = Very Severe
Time Frame: Change from baseline for month 2
Population: ITT with LOCF
Measure: Mean (Standard Deviation); unit: Scale score
Arm/Group | Lubiprostone Study Period I | Placebo Study Period I
Number analyzed (Participants) | 390 | 193
Scale score | -0.58 (0.846) | -0.43 (0.762)
Statistical Analysis 1: Comparison: Lubiprostone Study Period I vs Placebo Study Period I; Test type: Superiority or Other; p = 0.049, van Elteren nonparametric test; Adjusted for center

18. Secondary Outcome: Month 3 Bowel Straining Change From Baseline
Description: 0 = Absent,1 = Mild, 2 = Moderate, 3 = Severe, and 4 = Very Severe
Time Frame: Change from baseline for month 3
Measure: Mean (Standard Deviation); unit: Scale score
Arm/Group | Lubiprostone Study Period I | Placebo Study Period I
Number analyzed (Participants) | 390 | 193
Scale score | -0.56 (0.847) | -0.45 (0.760)
Statistical Analysis 1: Comparison: Lubiprostone Study Period I vs Placebo Study Period I; Test type: Superiority or Other; p = 0.348, van Elteren nonparametric test; Adjusted for center

19. Secondary Outcome: Month 2 Constipation Severity Change From Baseline
Description: 0 = Absent, 1 = Mild, 2 = Moderate, 3 = Severe, and 4 = Very Severe
Time Frame: Change from baseline for month 2
Population: ITT with LOCF
Measure: Mean (Standard Deviation); unit: Scale score
Arm/Group | Lubiprostone Study Period I | Placebo Study Period I
Number analyzed (Participants) | 390 | 193
Scale score | -0.50 (0.719) | -0.40 (0.670)
Statistical Analysis 1: Comparison: Lubiprostone Study Period I vs Placebo Study Period I; Test type: Superiority or Other; p = 0.064, van Elteren nonparametric test; Adjusted for center

20. Secondary Outcome: Month 3 Constipation Severity Change From Baseline
Description: 0 = Absent, 1 = Mild, 2 = Moderate, 3 = Severe, and 4 = Very Severe
Time Frame: Change from baseline for month 3
Population: ITT with LOCF
Measure: Mean (Standard Deviation); unit: Scale score
Arm/Group | Lubiprostone Study Period I | Placebo Study Period I
Number analyzed (Participants) | 390 | 193
Scale score | -0.51 (0.755) | -0.41 (0.712)
Statistical Analysis 1: Comparison: Lubiprostone Study Period I vs Placebo Study Period I; Test type: Superiority or Other; p = 0.111, van Elteren nonparametric test

21. Secondary Outcome: Month 2 Symptom Relief
Description: as for outcome 5
Time Frame: Change from baseline for month 2
Population: ITT with LOCF
Measure: Mean (Standard Deviation); unit: Scale score
Arm/Group | Lubiprostone Study Period I | Placebo Study Period I
Number analyzed (Participants) | 390 | 193
Scale score | 0.76 (1.278) | 0.59 (1.203)
Statistical Analysis 1: Comparison: Lubiprostone Study Period I vs Placebo Study Period I; Test type: Superiority or Other; p = 0.144, Cochran-Mantel-Haenszel; Stratified by pooled center

22. Secondary Outcome: Month 3 Symptom Relief
Description: as for outcome 5
Time Frame: Change from baseline for month 3
Population: ITT with LOCF
Measure: Mean (Standard Deviation); unit: Scale score
Arm/Group | Lubiprostone Study Period I | Placebo Study Period I
Number analyzed (Participants) | 390 | 193
Scale score | 0.74 (1.259) | 0.57 (1.277)
Statistical Analysis 1: Comparison: Lubiprostone Study Period I vs Placebo Study Period I; Test type: Superiority or Other; p = 0.168, Cochran-Mantel-Haenszel; Adjusted by pooled center

23. Secondary Outcome: Month 1 Abdominal Bloating Change From Baseline
Description: 0 = Absent, 1 = Mild, 2 = Moderate, 3 = Severe, and 4 = Very Severe
Time Frame: Change from baseline for month 1
Population: ITT with LOCF
Measure: Mean (Standard Deviation); unit: Scale score
Arm/Group | Lubiprostone Study Period I | Placebo Study Period I
Number analyzed (Participants) | 390 | 193
Scale score | -0.30 (0.585) | -0.24 (0.516)
Statistical Analysis 1: Comparison: Lubiprostone Study Period I vs Placebo Study Period I; Test type: Superiority or Other; p = 0.615, van Elteren nonparametic test; Adjusted for center

24. Secondary Outcome: Month 1 Bowel Movement Frequency Rates Change From Baseline
Time Frame: Change from baseline for month 1
Population: ITT, with LOCF
Measure: Mean (Standard Deviation); unit: BM/week
Arm/Group | Lubiprostone Study Period I | Placebo Study Period I
Number analyzed (Participants) | 390 | 193
BM/week | 1.22 (2.234) | 0.88 (2.093)
Statistical Analysis 1: Comparison: Lubiprostone Study Period I vs Placebo Study Period I; Test type: Superiority or Other; p = 0.108, van Elteren nonparametric test

25. Secondary Outcome: Month 2 Bowel Movement Frequency Rates Change From Baseline
Time Frame: Change from baseline for month 2
Population: ITT, with LOCF
Measure: Mean (Standard Deviation); unit: BM/week
Arm/Group | Lubiprostone Study Period I | Placebo Study Period I
Number analyzed (Participants) | 390 | 193
BM/week | 1.23 (2.440) | 1.10 (2.581)
Statistical Analysis 1: Comparison: Lubiprostone Study Period I vs Placebo Study Period I; Test type: Superiority or Other; p = 0.483, van Elteren nonparametric test

26. Secondary Outcome: Month 3 Bowel Movement Frequency Rates Change From Baseline
Time Frame: Change from baseline for month 3
Population: ITT, with LOCF
Measure: Mean (Standard Deviation); unit: BM/week
Arm/Group | Lubiprostone Study Period I | Placebo Study Period I
Number analyzed (Participants) | 390 | 193
BM/week | 1.15 (2.744) | 1.04 (2.731)
Statistical Analysis 1: Comparison: Lubiprostone Study Period I vs Placebo Study Period I; Test type: Superiority or Other; p = 0.491, van Elteren nonparametric test

27. Secondary Outcome: Month 1 Abdominal Pain Change From Baseline
Description: 0 = Absent, 1 = Mild, 2 = Moderate, 3 = Severe, and 4 = Very Severe
Time Frame: Change from baseline for month 1
Measure: Mean (Standard Deviation); unit: Scale Score
Arm/Group | Lubiprostone Study Period I | Placebo Study Period I
Number analyzed (Participants) | 390 | 193
Scale Score | -0.29 (0.588) | -0.27 (0.508)
Statistical Analysis 1: Comparison: Lubiprostone Study Period I vs Placebo Study Period I; Test type: Superiority or Other; p < 0.001, van Elteren nonparametric test; Adjusted for center

28. Secondary Outcome: Month 2 Abdominal Pain Change From Baseline
Description: 0 = Absent, 1 = Mild, 2 = Moderate, 3 = Severe, and 4 = Very Severe
Time Frame: Change from baseline for month 2
Measure: Mean (Standard Deviation); unit: Scale Score
Arm/Group | Lubiprostone Study Period I | Placebo Study Period I
Number analyzed (Participants) | 390 | 193
Scale Score | -0.43 (0.695) | -0.37 (0.614)
Statistical Analysis 1: Comparison: Lubiprostone Study Period I vs Placebo Study Period I; Test type: Superiority or Other; p < 0.001, van Elteren nonparametric test; Adjusted for center

29. Secondary Outcome: Month 3 Abdominal Pain Change From Baseline
Description: 0 = Absent, 1 = Mild, 2 = Moderate, 3 = Severe, and 4 = Very Severe
Time Frame: Change from baseline for month 3
Measure: Mean (Standard Deviation); unit: Scale Score
Arm/Group | Lubiprostone Study Period I | Placebo Study Period I
Number analyzed (Participants) | 390 | 193
Scale Score | -0.42 (0.722) | -0.36 (0.684)
Statistical Analysis 1: Comparison: Lubiprostone Study Period I vs Placebo Study Period I; Test type: Superiority or Other; p < 0.001, van Elteren nonparametric test; Adjusted for center

ADVERSE EVENTS:
Time Frame: Up to 12 weeks
Description: Any subject who took at least 1 dose of study medication made up the safety population. The N of this population is different from both the total subjects randomized and the ITT population
Groups:
- Lubiprostone Study Period I: 8 mcg capsules twice daily (BID)
- Placebo Study Period I: Matching placebo capsules twice daily (BID)
Arm/Group | Lubiprostone Study Period I | Placebo Study Period I
Serious Adverse Events (participants affected / at risk) | 5/396 | 2/192
Other Adverse Events (participants affected / at risk) | 75 | 25
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lubiprostone Study Period I (N=396) | Placebo Study Period I (N=192)
Thyroid gland cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Mitral valve incompetence (Cardiac disorders) | 1 (1) | 0 (0)
Coronary artery disease (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac arrest (Cardiac disorders) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0)
Dysuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Back injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected / at risk (number of events):
Term (organ system) | Lubiprostone Study Period I | Placebo Study Period I
Nausea (Gastrointestinal disorders) | 47/396 (47) | 11/192 (11)
Diarrhoea (Gastrointestinal disorders) | 28/396 (28) | 11/192 (11)
Abdominal Pain (Gastrointestinal disorders) | 22/396 (22) | 12/192 (12)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No